CLINICAL TRIAL: NCT02915094
Title: Kineret in the Treatment of Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: KIRA
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anakinra
  Other Names: Kineret

SUMMARY:
Objective of the study is to gain knowledge about the administration of Kineret in patients with rheumatoid arthritis in the daily routine treatment and not in controlled trials. In the current survey, the investigation of the response rate of Kineret regarding the date of onset of action, the efficacy, as well as the tolerability and safety are of particular interest.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the patient
* Rheumatoid arthritis
* Previous methotrexate therapy with inadequate response

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male and female patients with rheumatoid Arthritis who are treated with Kineret according to the therapeutic decision of the attending physician.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score 28 (DAS28) | 0-52 weeks
  The DAS28 measures the progress and improvement of Rheumatoid Arthritis. DAS28 values range from 2.0 to 10.0 while higher values mean a higher disease activity. A DAS 28 below the value of 2.6 is interpreted as Remission. Both the number of joints with tenderness upon touching and swelling are counted. In addition, the erythrocyte sedimentation rate is measured. Also, the patient makes a subjective assessment of disease activity during the preceding 7 days on a scale between 0 and 100, where 0 is "no activity" and 100 is "highest activity possible".
ACR response | 0-52 weeks
  The ACR (American College of Rheumatology) Criteria measures the effectiveness of treatments for Rheumatoid Arthritis. The ACR is reported as % improvement, comparing disease activity at two discrete time points.
Health Assessment Questionnaire | 0-52 weeks
  The patients will at each visit complete a questionnaire about their health status and the impairment in usual activities due to the rheumatoid disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zeitler, MD, Study Director — Swedish Orphan Biovitrum GmbH
Locations (1):
- Swedish Orphan Biovitrum Investigational Site, Freiburg im Breisgau, Germany